CLINICAL TRIAL: NCT03123393
Title: Phase 2 Study of TAK-659 in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma After at Least 2 Prior Lines of Chemotherapy
Brief Title: TAK-659 in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy of the drug; no safety concern
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C34004; U1111-1187-6208 (Other: WHO); 2016-003716-12 (EudraCT Number); 17/YH/0181 (Registry Identifier: NRES)
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Drug therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — TAK-659

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: TAK-659 100 mg (Experimental): TAK-659 100 mg tablet, orally, once daily (QD), during each 28-days cycle (median exposure was 41 days).
  Interventions: Drug: TAK-659
- Cohort B: TAK-659 Ramp-up Dosing (Experimental): TAK-659 60-100 mg tablet, orally, QD, dose based on safety and tolerability during each 28-days cycle (median exposure was 28 days).
  Interventions: Drug: TAK-659

INTERVENTIONS:
Drug: TAK-659 — TAK-659 Tablets

SUMMARY:
The purpose of this study is to assess the efficacy of TAK-659 measured by independent radiologic review committee (IRC)-assessed overall response rate (ORR) in participants with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
The drug being tested is TAK-659. This study will evaluate overall response rate (ORR) in participants with relapsed or refractory DLBCL who take TAK-659.

The study will enroll approximately 122 participants. Participants will be assigned to:

• TAK-659 60 mg to 100 mg

All participants will be asked to take the tablets of TAK-659 at the same time each day throughout the study in a 28-day cycle.

This multi-center trial will be conducted in the United States, United Kingdom, Spain, Italy, France, Canada, Germany. The overall time to participate in this study is approximately 48 months. Participants will be assessed for disease response and progression during the PFS follow-up every 3 months after end of treatment (for participants who discontinue due to reasons other than disease progression) and OS follow-up every 3 months from the last dose of study drug until death or conclusion of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Must have histologically confirmed DLBCL, including de novo disease or transformed disease from indolent NHL.

   a. High-grade B-cell lymphoma (BCL) with MYC and BCL-2 and/or BCL-6 translocations (double-hit DLBCL under DLBCL, not otherwise specified [NOS], based on the 2008 World Health Organization [WHO] classification criteria) is not eligible for this study.
2. Local pathology review for histological confirmation; A formalin-fixed, paraffin-embedded (FFPE) tumor block or appropriately stained slides from a fresh biopsy is required.
3. Relapsed or refractory to greater than or equal to (>=) 2 prior lines of chemotherapy based on standard of care with certain requirements for prior therapy.
4. Documented investigator-assessed relapse or progression after the last treatment is required if the participant responded and then progressed on the prior treatment.
5. Measurable disease per IWG 2007 criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status less than (<) 2.
7. Life expectancy of greater than (>) 3 months.
8. Adequate organ function, including the following:

   1. Bone marrow reserve: absolute neutrophil count (ANC) >=1000/microliter (μL), platelet count >=75,000/μL (>=50,000/μL for participants with bone marrow involvement), and hemoglobin >=8 gram per deciliter (g/dL).
   2. Hepatic: total bilirubin less than or equal to (<=) 1.5 times the upper limit of the normal range (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.5*ULN.
   3. Renal: creatinine clearance >=60 milliliter per minute (mL/min).
   4. Others:

      * Lipase <=1.5*ULN and amylase <=1.5*ULN with no clinical symptoms suggestive of pancreatitis or cholecystitis.
      * Blood pressure <=Grade 1 (hypertensive participants are permitted if their blood pressure is controlled to <=Grade 1 by hypertensive medications.
      * Glycosylated hemoglobin is <=6.5% hyperglycemic participants permitted if glucose is well controlled by antihyperglycemic medication).

Exclusion Criteria:

1. Central nervous system (CNS) lymphoma; active brain or leptomeningeal metastases.
2. Known human immunodeficiency virus (HIV)-related malignancy.
3. Systemic anticancer treatment (including investigational agents) less than 3 weeks before the first dose of study treatment (<=4 weeks for antibody-based therapy including unconjugated antibody, antibody-drug conjugate, and bi-specific T-cell engager agents; <=8 weeks for cell-based therapy or anti-tumor vaccine).
4. Radiotherapy less than 3 weeks before the first dose of study treatment. If prior radiotherapy occurred <4 to 6 weeks before study start, as radiated lesions cannot be reliably assessed by fluorodeoxyglucose-positron emission tomography (FDG-PET), nonradiated target lesions are required for eligibility, and prior radiotherapy information must be submitted to the IRC.
5. Known HIV positive, hepatitis B surface antigen positive or known or suspected active hepatitis C infection.
6. Prior autologous stem cell transplant (ASCT) within 6 months or prior ASCT at any time without full hematopoietic recovery before Cycle 1 Day 1, or allogeneic stem cell transplant any time.
7. Participants with certain cardiovascular conditions are excluded.
8. Major surgery within 14 days before the first dose of study drug or incomplete recovery from any complications from surgery.
9. Systemic infection requiring parenteral antibiotic therapy or other serious infection (bacterial, fungal, or viral) within 21 days before the first dose of study drug.
10. Treatment with high-dose corticosteroids for anticancer purposes within 7 days before the first dose of TAK-659.
11. Participants with another malignancy within 2 years of study start. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection and are considered disease-free at the time of study entry.
12. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659.
13. Received medications, supplements, or food/beverages that are P-glycoprotein (P-gp) inhibitors or inducers or strong cytochrome P450 (CYP) 3A inhibitors or inducers within a certain timeframe prior to the first dose of study drug. Depending on the substance, the washout period for P-gp inhibitors or inducers or strong CYP3A inhibitors or inducers will be either 7 days or 5 times the half-life (half-life is related to the time required for elimination from the body). The washout period for grapefruit containing food or beverages is 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (41):
- United States (10):
  - University of Kansas Medical Center, Westwood, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Swedish Medical Oncology - Edmonds, Edmonds, Washington
  - Swedish Cancer Institute - Issaquah, Issaquah, Washington
  - Swedish Health Services, Seattle, Washington
  - University of Washington, Hutchinson Cancer Research Center, Seattle, Washington
  - Swedish First Hill Campus, Seattle, Washington
- Canada (3):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - CHU de Quebec -Universite Laval-Hopital de L'Enfant Jesus, Québec, Quebec
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
- France (10):
  - Hopital Haut-Leveque, Pessac, Aquitaine
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHRU Clermont- Ferrand CHU Estaing, Clermont-Ferrand, Auvergne
  - Centre Henri-Becquerel, Rouen, Haute-normandie
  - Hopital Dupuytren, Limoges, Limousin, Lorraine
  - Institut Paoli Calmettes Departement de Recherche Clinique et de l'Innovation, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hopital Necker-Enfants Malades, Paris, Île-de-France Region
  - Hopital Saint Louis, Paris, Île-de-France Region
  - Groupe Hospitalier - Hopitaux Universitaires Pitie-Salpetriere - Charles-Foix - Pitie-Salpetriere, Paris, Île-de-France Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Italy (6):
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero-Universitaria "Maggiore della Carita", Novara
  - Azienda Ospedaliero Universitaria Santa Maria della Misericordia di Udine, Udine
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario La Fe, Valencia
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham, England
  - London North West Healthcare NHS Trust, Imperial College London, Harrow, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne, England

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 26 investigative sites in France, Great Britain, Italy, Spain, Canada, United States from 10 October 2017 to 17 December 2019. The study was terminated by the sponsor before the initiation of the stage 2 efficacy evaluation.
Pre-assignment Details: Participants with a diagnosis of relapsed or refractory diffuse large B-cell lymphoma who had at least 2 prior lines of chemotherapy were enrolled in Cohorts A and B. Cohort A received a single dose and Cohort B received ramp-up doses of TAK-659 in Stage 1 of the study.
Period: Overall Study
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Started | 24 | 25
Completed | 3 | 2
Not Completed | 21 | 23
Not completed — Study Terminated by Sponsor | 6 | 9
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Reason not Specified | 13 | 13

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of TAK-659.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.01) | 64.6 (11.37) | 64.4 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 18 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Non-Hispanic and Latino | 21 | 13 | 34
  Not Reported | 2 | 7 | 9
  Unknown | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  France | 3 | 11 | 14
  United Kingdom | 3 | 3 | 6
  Italy | 4 | 4 | 8
  Spain | 3 | 3 | 6
  Canada | 1 | 0 | 1
  United States | 10 | 4 | 14
Height [Mean (Standard Deviation); unit: cm] | 172.8 (9.55) | 167.5 (9.52) | 170.1 (9.81)
Weight [Mean (Standard Deviation); unit: kg] | 92.88 (21.132) | 72.81 (18.388) | 82.64 (22.040)

OUTCOME MEASURES:

1. Primary Outcome: Stage 2: ORR as Assessed by Independent Radiologic Review Committee (IRRC) Based on Modified 2007 International Working Group (IWG) Criteria
Description: ORR was defined as the percentage of participants with complete response (CR), or partial response (PR) as assessed by IRRC according to the modified 2007 IWG criteria for malignant lymphoma. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Stage 2: CR Rate as Assessed by IRC Based on Modified 2007 IWG Criteria
Description: CR rate was defined as percentage of participants with complete response as assessed by IRC according to the modified 2007 IWG. CR was defined as disappearance of all evidence of disease.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Stage 2: ORR as Assessed by IRRC Based on 2014 IWG-Lugano Criteria
Description: ORR was defined as the percentage of participants with CR or PR as assessed by IRRC according to the 2014 Lugano classification, IWG criteria for malignant lymphoma. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Stage 2: CR Rate as Assessed by IRRC Based on 2014 IWG-Lugano Criteria
Description: CR rate was defined as percentage of participants with complete response as assessed by IRC according to the 2014 Lugano classification, IWG criteria. CR was defined as disappearance of all evidence of disease.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Stage 2: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a CR/PR to the date of first documentation of tumor progression or progressive disease (PD) per IRRC assessment according to IWG criteria. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites. PD was defined as presence of any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Stage 2: Duration of CR
Description: Duration of CR was defined as the time from the date of first documentation of a CR/PR to the date of first documentation of tumor progression or PD per IRRC assessment according to IWG criteria. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites. PD was defined as presence of any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Stage 2: ORR as Assessed by IRRC in Participants With Germinal Center B-cell (GCB) DLBCL
Description: ORR was defined as the percentage of participants with CR or PR as assessed by IRRC according to the modified 2007 IWG criteria for malignant lymphoma. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Stage 2: ORR as Assessed by IRC in Participants With DLBCL Transformed From Indolent Non-Hodgkin's Lymphoma (NHL)
Description: ORR was defined as the percentage of participants with CR or PR as assessed by IRC according to the modified 2007 IWG criteria for malignant lymphoma. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites.
Time Frame: Up to 12 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Stage 2: Progression Free Survival (PFS) as Assessed by IRC
Description: PFS was defined as time from start of study treatment to first documentation of PD per IRC assessment or up to death due to any cause, whichever occurs first based on IWG criteria. PD was defined as presence of any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: Up to 18 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Stage 2: Overall Survival (OS)
Description: OS was defined as the time from start of study treatment to date of death due to any cause.
Time Frame: Up to 24 months
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Stage 1: ORR as Assessed by IRRC to Select Stage 2 Dose Regimen of TAK-659 From the Lead-in Dose Exploration Phase
Description: ORR was defined as the percentage of participants with CR or PR as assessed by IRC. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites.
Time Frame: Up to 12 months
Population: Data were not reported for this outcome measure because ORR was only assessed by the investigator on this study and not by IRRC as the study was terminated and the selection of dose for Stage 2 was not applicable.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Stage 2: ORR as Assessed by IRC at 3, 6, and 9 Cycles in Participants With DLBCL
Description: as for outcome 8
Time Frame: At Cycles 3, 6 and 9 (Up to 12 months) (Each cycle of 28 days)
Population: As the study was terminated before the initiation of Stage 2, data was not collected for this outcome measure.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent form (ICF) through 28 days after administration of the last dose of study drug or until the start of subsequent anticancer therapy, whichever occurs first (Up to approximately 14 months).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort A: TAK-659 100 mg | Cohort B: TAK-659 Ramp-up Dosing
All-Cause Mortality (participants affected / at risk) | 3/24 | 3/25
Serious Adverse Events (participants affected / at risk) | 14/24 | 13/25
Other Adverse Events (participants affected / at risk) | 24/24 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: TAK-659 100 mg (N=24) | Cohort B: TAK-659 Ramp-up Dosing (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Lymphocytic infiltration (Blood and lymphatic system disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Asthenia (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Enterovirus infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pulmonary nocardiosis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: TAK-659 100 mg (N=24) | Cohort B: TAK-659 Ramp-up Dosing (N=25)
Fatigue (General disorders) | 6 | 8
Oedema peripheral (General disorders) | 7 | 2
Asthenia (General disorders) | 3 | 1
Oedema (General disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 5
Alanine aminotransferase increased (Investigations) | 7 | 4
Amylase increased (Investigations) | 6 | 4
Blood creatine phosphokinase increased (Investigations) | 6 | 2
Lipase increased (Investigations) | 4 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 4 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 2
C-reactive protein increased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Periorbital oedema (Eye disorders) | 5 | 3
Vision blurred (Eye disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Oral candidiasis (Infections and infestations) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Hypertension (Vascular disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Pyrexia (General disorders) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT03123393/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03123393/SAP_001.pdf